CLINICAL TRIAL: NCT07162233
Title: Assessment and Maintenance of Derotation Osteotomy Utilizing Kirschner Wires for the Correction of Congenital Proximal Radioulnar Synostosis
Brief Title: Surgical Corection of Congenital Proximal Radioulnar Synostosis Using Double Osteotomy Technique.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Refaat Mohamed Hassan, Assessment and maintenance of derotation osteotomy utilizing Kirschner wires for the correction of congenital proximal radioulnar synostosis, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med--25-8-4MS
Record Dates: First submitted 2025-08-30; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Synostosis
MeSH Terms: conditions — Synostosis

STUDY DESIGN:
Intervention Model Description: The aim of the work is to asses and maintain derotation osteotomy for treating proximal radioulnar synostosis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- child 4 : 12 age with congenital radioulnar synostosis (Experimental): Assessment and maintenance of derotation osteotomy utilizing Kirschner wires for the correction of congenital proximal radioulnar synostosis
  Interventions: Procedure: derotation osteotomy utilizing Kirschner wires for the correction of congenital proximal radioulnar synostosis

INTERVENTIONS:
Procedure: derotation osteotomy utilizing Kirschner wires for the correction of congenital proximal radioulnar synostosis — The level of distal radial and proximal ulnar osteotomies is determined under C- arm. A k-wire is inserted in the outer border of the metaphysis of the radius distal to the level of the osteotomy, engaging and transfixing the radioulnar joint, small skin incision is made over the dorsal aspect of the forearm at the level of distal radial osteotomy, dissection of subcutaneous tissue with good exposure of the extensor tendons, transverse osteotomy is done using 2.5 mm drill bit and small sharp osteotme, allowing derotation movement of the distal part of the radius using the k-wire.
  Another small skin incision is made over the level of proximal ulnar osteotomy, dissection of subcutaneous tissue, another ulnar transverse osteotomy is done distal to the level of the proximal radioulnar synostosis. Derotaion of the forearm is adjusted in the functional position of the forearm in around (10˚:20˚supination), wound closure using absorbable Vicryl sutures. Above elbow cast is used f

SUMMARY:
The purpose of the present study is to asses and maintain derotation osteotomy for treating proximal radioulnar synostosis.

DETAILED DESCRIPTION:
Proximal radio-ulnar synostosis is a skeletal malformation of the up-per limb characterized by bony fusion at the proximal aspect of the radius and ulna. The proximal third is considered the most common site of the radio-ulnar synostosis.

Congenital proximal radioulnar synostosis is an uncommon genetic malformation of the upper limb.

This deformity is found mainly in preschool-aged children (4:8 years old), The proximal radioulnar synostosis was first described by the Dutch anatomist Eduard Sandifort in 1793¹.

Although Congenital radio ulnar synostis is an uncommon congenital disease, it is the most common congenital disorder affecting the elbow and forearm joint ,being bilateral in 60-80% of cases .

there is no gold standard option for the treatment of congenital proximal radioulnar synostosis. The ideal treatment for congenital radioulnar synostosis aims to restore rotational function and prevents the recurrence of the bony bridges. Both conservative and surgical treatments are possible, but results are still controversial, the main indication for surgical treatment is the limitation of daily activities. Many surgical methods have been reported aiming restoration of radius rotation around the ulna such as Synostosis resection and artificial bio-logical tissue interposition and derotational osteotomies².

Historically, surgical separation of the synostosis and vascularized and non-vascularized interposition techniques to fill the interosseous space and prevent scar formation and resynostosis had theoretically been considered the ideal treatment³. Nowdays, the leading methods of surgical treatment of Congenital radio ulnar synostosis are precisely the variants of forearm derotation osteotomies such as : gradual correction of pronation deformity using external fixation devices , performing a single-level osteotomy of the radius , osteoto-my of both forearm bones at different levels and osteotomy through the synostosis zone⁴.

ELIGIBILITY:
Inclusion Criteria:

* Patients with congenital idiopathic proximal radioulnar synostosis at the age of 4:12 years old.

Exclusion Criteria:

* patients with post traumatic proximal radioulnar synostosis, patients with distal ra-dioulnar synostosis and patients with neuromuscular disorder.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
surgical derotation osteotomy utilizing Kirschner wires for the correction of congenital proximal radioulnar synostosis | one year
  Proximal radio-ulnar synostosis is a skeletal malformation of the upper limb characterized by bony fusion at the proximal aspect of the radius and ulna. The proximal third is considered the most common site of the radio-ulnar synostosis.
  This deformity is found mainly in preschool-aged children (4:8 years old), The proximal radioulnar synostosis was first described by the Dutch anatomist Eduard Sandifort in 1793¹.
  The ideal treatment for congenital radioulnar synostosis aims to restore rotational function and prevents the recurrence of the bony bridges. we aim to do surgical osteotomy and correct the synostosis to restore the function of the upper limb and will be assessed by geniometry , clinical and functional outcomes .

CONTACTS AND LOCATIONS:
Overall Officials: Marwan shams eldeen, MD orthopedeic, Study Chair — Sohag University
Locations (1):
- Sohag Faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR